CLINICAL TRIAL: NCT05812170
Title: Awareness, Control and Treatment of Urinary Incontinence and Other Pelvic Floor Dysfunctions in Female Athletes
Brief Title: Pelvic Floor Dysfunctions and Female Athletes
Acronym: ACTITUD1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: Fundació d'investigació Sanitària de les Illes Balears (Other Government); Consejo Superior de Deportes, Spain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 124CER19
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-03

CONDITIONS: Pelvic Floor Disorders
Keywords: Female; Athlete; Track and Field; Education
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: A quasiexperimental controlled trial is designed, with two arms: an experimental group and a control group.
Masking Description: The design of this study does not allow to mask participants, care providers, investigators or outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Educational online session about PF (Experimental): Participants will attend an 90-minutes educational online session.
  Interventions: Behavioral: Educational online session about PF
- Control (No Intervention): Despite the fact that all athletes will be invited to participate in the study, those who did not attend the educational session will be considered as control group. These participants will not receive any educational session or information about PF prior to be evaluated.

INTERVENTIONS:
Behavioral: Educational online session about PF — The educational online session will last 90 minutes, as follows: 10 minutes of contextualization, 40 minutes of practical content about pelvic floor consciousness and 40 of theoretical content (anatomy and practices related to PFD).
  Arms: Educational online session about PF

SUMMARY:
Pelvic floor dysfunctions (PFD) are especially prevalent among females athletes due to the efforts from sports practice. As conservational management, increasing the athletes' information regard important research lines. However, embarrassment of female athletes limits educational or health demands and facilitate an invisible condition, potentially influenced by gender stereotypes. New technologies could facilitate engaging virtual educational approaches. This study will evaluate the effects of an educational online session about PFD in the knowledge about it, and practices related with it, existing gender stereotypes and PFD diagnosis of female athletes. To this end, all female athletes who practice Track and Field in Spain will be invited to attend an educational online session with theoretical-practical content about PF. As eligibility criteria, participants should train and compete in any of the Track and Field modalities, and have federative license from regional or national Track and Field Federation at the moment of the start of the study. Participants should have at least 18 years old. The investigators expect 400 athletes to fulfill the questionnaires, of which the investigators expect 200 to attend the educational online session.

Before the educational online session, all female athletes will reply an anonymous questionnaire to inform about their knowledge of PFD, daily practices related to PFD, influencing gender stereotypes and PFD auto-reported diagnosis. One month later, this questionnaire will be sent to female athletes (both athletes who attended the educational session or not) to describe changes after attending the online educational session and compared to those athletes who did not attend it. The main outcomes will be the level of knowledge about PF, the number of detrimental practices potentially related to PFD, the number of healthy practices to care PF and existence of influencing gender stereotypes. As an additional outcome, it will be considered the PFD auto-reported diagnosis.

DETAILED DESCRIPTION:
The educational online session will last 90 minutes, as follows: 10 minutes of contextualization, 40 minutes of practical content about pelvic floor consciousness and 40 of theoretical content (anatomy and practices related to PFD). Also, a 3D realistic virtual model of pelvic floor structures will be used.

ELIGIBILITY:
Inclusion Criteria:

* To train and compete in any of the Track and Field modalities
* To have federative license from regional or national Track and Field Federation in the season when study starts.

Exclusion Criteria:

* Non-applicable

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 281 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Knowledge about pelvic floor | One month
  Change in the level of knowledge about PF according to the responses to online questionnaire after attending the online educational session and compared to those athletes who do not attend educational session. To assess it, participants will reply an ad-hoc questionnaire with ten multiple-choice questions about pelvic floor structures. It will be counted the number of correct answers (0 points as the worst punctuation, 10 points as the best punctuation).
Detrimental practices related to pelvic floor dysfunctions | One month
  Change in number of detrimental practices that participants often carry out during their daily life, potentially related to pelvic floor dysfunctions, after attending the online educational session and compared to those athletes who do not attend educational session.
Healthy practices to care pelvic floor | One month
  Change in number of healthy practices to care pelvic floor that participants often carry out during their daily life, after attending the online educational session and compared to those athletes who do not attend educational session.

SECONDARY OUTCOMES:
Gender stereotypes | One month
  Change in number of existing gender stereotypes that potentially influence PFD, after attending the online educational session and compared to those athletes who do not attend educational session.
PFD auto-reported diagnosis | One month
  It will be considered if PFD is auto-reported through the questionnaire that athletes will reply. To this end, athletes will reply five yes-no questions regarding the existence of PFD. In case of affirmative response in any of these diagnostic questions by an athlete, it will be considered that this athlete has a PFD. Between-group differences were considered.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Romero-Franco, PhD, Principal Investigator — University of the Balearic Islands
Locations (1):
- University of the Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No